## Statistical analysis plan

The data are presented as means with standard deviations (SD), medians with interquartile range (IQR) or counts with percentages. Results were analyzed by the Chisquare test, Mann–Whitney U test and by Fisher's exact test. p values less than 0.05 were considered to be statistically significant. Univariable logistic regression analysis with beta coefficient and 95% confidence intervals (95% CIs) was used to assess risk factors for high radiation dose and fluoroscopy time. A logarithmic transformation was performed with the KAP and FT due to asymmetrical distribution. Statistical analyses were carried out using SPSS statistical software, version 24 (SPSS, Inc., Chicago, IL, USA).